CLINICAL TRIAL: NCT05573425
Title: Comparing the Efficacy of Topical Tazarotene Gel 0.1% Versus Microneedling in Atrophic Post Acne Scars
Brief Title: Comparing the Efficacy of Topical Tazarotene Gel 0.1% v/s Microneedling in Atrophic Post Acne Scars
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr Faiza Shabbir, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jpmc
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Acne Scar
Keywords: Tazarotene
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group on Treatment:Tazarotene Gel (Active Comparator): In group A, patients were instructed to apply a thin film of tazarotene gel 0.1% over the affected area once daily in the evening by placing a pea-sized amount of gel in the palm of the hand and using tip of a finger to cover the entire half of the face. Patients who experienced facial dryness were allowed to use a moisturizing cream during the day on entire face but use of any other medication on the face was prohibited.
  Intervention - Tazarotene gel 0.1%
  Interventions: Drug: Tazarotene gel 0.1%
- Group on Treatment:Microneedling (Active Comparator): In group B, microneedling was performed with a standard dermaroller (192 needles of length 1.5 mm) by the same investigator, once per month for 6 months. A topical anesthetic mixture of lignocaine and prilocaine was applied over the face in a thick layer under occlusion 1 hour before the procedure.
  Microneedling was performed by rolling the dermaroller with uniform and firm pressure in 4 different directions (i.e, perpendicular and diagonal to each other) with to-and-fro motion up to 8 times (a total of 32 passes) or until the end point of uniform pinpoint bleeding was achieved. After treatment, the area was wetted with saline pads. The participants were instructed to follow strict photoprotective measures including the application of a broad-spectrum sunscreen with sun protection factor 30 over the entire face.
  Intervention - Microneedling via dermarolller
  Interventions: Device: Microneedling

INTERVENTIONS:
Drug: Tazarotene gel 0.1% — Tazarotene gel 0.1% applied daily on Acne Scars.
  Other Names: Tazret gel 0.1%
  Arms: Group on Treatment:Tazarotene Gel
Device: Microneedling — Microneedling via dermaroller device performed on Acne Scars monthly.
  Other Names: Dermaroller device
  Arms: Group on Treatment:Microneedling

SUMMARY:
The purpose of this study was to compare the Efficacy of Topical Tazarotene gel 0.1% versus Microneedling in atrophic Post acne scars. All patients of age 18-40 years, with grade 2 to grade 4 facial atrophic acne scars, assessed using the Goodman and Baron qualitative global scarring grading. Group A was given daily home application of Topical Tazarotene gel 0.1% while on Group B, Microneedling monthly sessions done for 12 weeks. The results were assessed by photographs, Goodman and Baron Qualitative Acne Scars Grading system at the start and end of treatment. SPSS 21 was used for data analysis which showed comparable efficacy of daily home based application of Topical Tazarotene gel 0.1% versus Microneedling monthly sessions in Atrophic Post Acne Scars.

DETAILED DESCRIPTION:
This was a randomized Control Trial, done in Department of Dermatology, Jinnah Postgraduate Medical Centre (JPMC), Karachi from August 22, 2020 to February 21, 2021.

A total of 202 patients with 101 in each group. The sample size was estimated using WHO sample size calculator using statistics for efficacy in topical Tazarotene gel (group A) as 30.5% and micro-needling (group B) as 47.2%,80% power of test and 95% confidence level. Both genders, 18 to 40 years with atrophic post-acne scar patients of duration 4 to 8 years were included. Informed consent was obtained. Patients with grade 2 to 4 facial atrophic post-acne scars assessed by Goodman and Baron qualitative global scarring grading system. While excluded pregnant/lactating woman, any prior allergy to given drug, history of keloidal tendency/hypertrophic scarring, active acne or acne marks such as red, black or brown macular marks, previous dermabrasion, laser resurfacing on face, facial scar due to reasons other than acne, collagen vascular disease, bleeding disorders, treatment history of <4 weeks for topical retinoid, alpha/beta hydroxyl acids, <3 months for microdermabrasion and <6 months for oral retinoids.

This study was conducted after approval from ethical review committee and CPSP. During the patient first visit, baseline photographs were captured with informed consent. Dermoscopic examinations of predominant scar type (such as icepick, rolling or boxcar) and the ssca severity assessed according to the Goodman and Baron qualitative acne scarring grading systems for every patient. All patients were randomly divided into two groups using computer-generated sequential number placed in sealed envelopes and opened only before the commencement of the study. In group A, patients were instructed to apply a thin film of tazarotene gel 0.1% over the affected area once daily in the evening by placing a pea-sized amount of gel in the palm of the hand and using tip of a finger to cover the entire half of the face. Patients who experienced facial dryness were allowed to use a moisturizing cream during the day on entire face but use of any other medication on the face was prohibited. In group B, microneedling was performed with a standard dermaroller (192 needles of length 1.5 mm) by the same investigator, once per month for 6 months. A topical anesthetic mixture of lignocaine and prilocaine was applied over the face in a thick layer under occlusion 1 hour before the procedure.

Microneedling was performed by rolling the dermaroller with uniform and firm pressure in 4 different directions (i.e, perpendicular and diagonal to each other) with to-and-fro motion up to 8 times (a total of 32 passes) or until the end point of uniform pinpoint bleeding was achieved. After treatment, the area was wetted with saline pads. The participants were instructed to follow strict photoprotective measures including the application of a broad-spectrum sunscreen with sun protection factor 30 over the entire face. All patients were followed up at 3 month and on 6 month from the baseline visit. Digital photographs were captured at 3 and 6 month follow-up visits. An improvement by 2 qualitative grades was considered excellent, by 1 grade was rated good, and by 0 grade was labeled a poor response. The outcome was the change from baseline in acne scar severity grade at 3 and 6 month follow-up visits. All the data was entered in a predesigned proforma. Biasness and confounder were controlled by strictly following the inclusion criteria.

SPSS version 21 was used for data compilation and analysis. Frequencies and percentages were computed for qualitative variables like gender, scar type, treatment, scar severity grade at baseline, after 3 and 6 months and efficacy. Quantitative variables were presented as mean ± SD like age and duration of acne. Comparison between both groups for efficacy was done by using Chi square test. Effect modifier like age, gender and duration of disease were controlled through stratification. Post stratification, Chi square test was applied for categorical variables. Consider P <0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age from 18 to 40 years.
* Atrophic post-acne scar patients with duration 4 to 8 years.
* Informed consent will be obtained.
* Patients with grade 2 to 4 facial atrophic post-acne scars as assessed by the Goodman and Baron qualitative global scarring grading system.

Exclusion Criteria:

* Pregnant or lactating woman.
* Patients having any allergy related to given drug.
* History of keloidal tendency or hypertrophic scarring.
* Those with active acne or acne marks such as red, black or brown macular marks.
* Patients with a previous history of dermabrasion or laser resurfacing on the face.
* Facial scar due to reasons other than acne, collagen vascular disease or bleeding disorder.
* Patients with a treatment history of <4 weeks for topical retinoid and alpha/beta hydroxy acids, <3 months for microdermabrasion and <6 months for oral retinoids.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Change in morphology of Acne Scars | 12 weeks
  There is a change in Acne Scars assessed by Goodman and Baron Qualitative Acne Scars Grading system

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, Study Director — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah Post graduate medical center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT05573425/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT05573425/ICF_001.pdf